CLINICAL TRIAL: NCT06779942
Title: FROG-ARDS: Correlation of IL-17A to Hyperinflammatory Biomarkers, Sub-phenotype, and Clinical Outcomes in Patients With Acute Respiratory Distress Syndrome in the FROG ICU Dataset
Brief Title: The Association Between IL17, Acute Respiratory Distress Syndrome and Acute Respiratory Failure
Acronym: FROG-ARDS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22920
Record Dates: First submitted 2025-01-07; First posted 2025-01-17 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Acute Respiratory Failure (ARF)
Keywords: Acute respiratory distress syndrome (ARDS); Acute Respiratory Failure (ARF); IL-17 Inhibitor
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Respiratory Distress Syndrome (ARDS): The index date is the date of diagnosis of ARDS. The patients will be followed from the index date until the outcome, death, or end of follow-up whichever comes first. This study builds on data from FROG ICU registry, which is an observational, prospective, multicenter cohort study. The evaluation of each patient is performed through a comprehensive clinical assessment, instrumental tests (electrocardiogram, echocardiogram) and biological parameters. All the data are collected at admission, during the stay as well as at discharge and in addition these patients are followed up for long-term outcomes after ICU discharge. This allows us to evaluate the effect of different biomarkers as well as level of care in the ICU on long-term outcomes.
  Patient Identification period: Aug 2011 - Jun 2013 Exposure window: ICU admission to discharge
- Acute Respiratory Failure (ARF): The index date is the date of diagnosis of ARF. The patients will be followed from the index date until the outcome, death, or end of follow-up whichever comes first. This study builds on data from FROG ICU registry, which is an observational, prospective, multicenter cohort study. The evaluation of each patient is performed through a comprehensive clinical assessment, instrumental tests (electrocardiogram, echocardiogram) and biological parameters. All the data are collected at admission, during the stay as well as at discharge and in addition these patients are followed up for long-term outcomes after ICU discharge. This allows us to evaluate the effect of different biomarkers as well as level of care in the ICU on long-term outcomes.
  Patient Identification period: Aug 2011 - Jun 2013 Exposure window: ICU admission to discharge

SUMMARY:
This study will look at a protein called Interleukin (IL)-17A and how it relates to health markers in patients with a serious lung condition known as Acute Respiratory Distress Syndrome (ARDS). IL-17A is part of the immune system and helps the body fight infections, but too much of it can lead to inflammation, which can be harmful.

The researchers want to find out if the levels of IL-17A in the blood are connected to important health outcomes for patients, such as whether they survive in the Intensive Care Unit (ICU), after 30 days, and after 60 days. They will also check how long patients can stay off a ventilator and how many days they need to use a mechanical ventilator. A ventilator is a machine that helps people breathe when their lungs are not working well.

In addition to the main goal, the researchers will study how IL-17A relates to a severe form of ARDS called the hyperinflammatory sub-phenotype. They will also look at how IL-17A connects with other health markers, including IL-6, soluble tumor necrosis factor receptor (sTNFR), IL8, Tumor Necrosis Factor (TNF)a, IL1beta, and IL23. These markers can give information about inflammation and how the body is responding to illness.

To compare results, the researchers will include a control group of patients who had Acute Respiratory Failure (ARF) but did not have ARDS. This control group will help them understand the differences between the two conditions.

This research will use data from the FROG-ICU Registry, which gathers information on patients in intensive care units across Europe. The registry tracks patients' health after they leave the ICU, focusing on the risk factors for death in the year following their discharge. The data comes from 28 different ICUs in 19 hospitals.

The researchers will create two groups of patients based on their diagnoses: one group with ARDS and another with ARF. By studying these groups, they hope to learn more about the role of IL-17A in ARDS and its potential impact on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* invasive mechanical ventilation support for at least 24 h and/or treatment with a positive inotropic agent (except dopamine) for more than 24 h
* ARDS patients:

  o Diagnosis of ARDS at the time of study inclusion and within 24-48 hours of bio sample collection
* ARF patients o Diagnosis of Acute respiratory Failure (ARF) who do not have sepsis at the time of study inclusion and within 24-48 hours of bio sample collection

Exclusion Criteria:

o Patients with ARF who later develop ARDS after the 24-48 hour bio sample draw time period will be excluded as they will not have had baseline bio samples drawn in relation to onset of ARDS.

* Patients less than 18 years old
* severe head injury (initial Glasgow Coma Scale < 8) or brain death or a persistent vegetative state
* pregnancy or breastfeeding
* transplantation in the past 12 months; not expected to survive or to leave the hospital
* no social security coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Using the data from FROG ICU registry, we will create two cohorts of patients using diagnosis codes:
  Acute Respiratory Distress Syndrome (ARDS) Acute Respiratory Failure (ARF) The FROG ICU registry is a completed, prospective, observational, multicenter cohort study, designed to assess the incidence and to identify the risk factors of all-cause mortality during the year following discharge from the ICU. Our study will retrospectively analyze this prospectively collected data.
  The evaluation of each patient is performed through a comprehensive clinical assessment, instrumental tests (electrocardiogram, echocardiogram) and biological parameters. All the data are collected at admission, during the stay as well as at discharge and in addition these patients are followed up for long-term outcomes after ICU discharge. This allows us to evaluate the effect of different biomarkers as well as level of care in the ICU on long-term outcomes.
Sampling Method: Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
ICU Mortality | Baseline to ICU discharge (at least 24h) or death
  Evaluate the association between Interleukin (IL)-17A level and mortality at the Intensive Care Unit (ICU) in patients with ARDS
30 Day Mortality | Baseline to 30 days after ICU admission or death
  Evaluate the association between IL-17A level and 30 Day mortality in patients with ARDS
60 Day Mortality | Baseline to 60 days after ICU admission or death
  Evaluate the association between IL-17A level and 60 Day mortality in patients with ARDS
Ventilator free survival | From baseline to ICU discharge, but at least for 24 hrs
  Evaluate the association between IL-17A level and ventilator free survival in patients with ARDS
Number of days on mechanical ventilator | From baseline to ICU discharge, but at least for 24 hrs
  Evaluate the association between IL-17A level and days on mechanical ventilator in patients with ARDS

SECONDARY OUTCOMES:
Hyperinflammatory ARDS subtype correlation | From baseline to ICU discharge, but at least for 24 hrs
  Evaluate the association between IL-17A and hyperinflammatory sub-phenotype of ARDS
Biomarker Correlation with IL-17A | From baseline to ICU discharge, but at least for 24 hrs
  Evaluate the correlation between IL-17A and multiple biomarkers including IL-6, sTNFR, IL8, Tumour Necrosis Factor (TNF)a, IL1beta, IL23 in patients with ARDS
Comparison of associated biomarkers in hypo-inflammatory phenotype of ARDS | From baseline to ICU discharge, but at least for 24 hrs
  Compare these associations with the association with these biomarkers in hypo-inflammatory phenotype of ARDS
Comparison of associated biomarkers in hyper and hypo-inflammatory phenotypes of Acute Respiratory Failure (ARF) | From baseline to ICU discharge, but at least for 24 hrs
  Compare these associations with the association with these biomarkers in the hyper and hypo-inflammatory phenotypes of Acute Respiratory Failure (ARF)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Saint Louis, Paris
  - University Paris Diderot, Paris

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Related Info — https://clinicaltrials.bayer.com/study/22920